CLINICAL TRIAL: NCT06677970
Title: Outcome in Patients Treated With Endovascular Thrombectomy - optIMAL Blood Pressure Control 2 (OPTIMAL-BP 2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2024-0880
Record Dates: First submitted 2024-09-23; First posted 2024-11-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Blood pressure; Ischemic stroke; thrombectomy; outcome
MeSH Terms: conditions — Ischemic Stroke | interventions — Nicardipine; Labetalol; urapidil; Phenylephrine

STUDY DESIGN:
Intervention Model Description: a multicenter, randomized, open Lable, blinded end-point clinical trial.
Who Masked: Outcomes Assessor
Masking Description: The mRS scores and adverse events were determined in participants at 1 month and 3 months via telephone or in person by local certified medical staff who were blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional BP magnagement group (SBP ≤180 mmHg) (Active Comparator)
  Interventions: Drug: BP lowering drugs (nicardipine, labetalol, urapidil)
- Intensive BP raising group (20% increase in SBP, maximum of 160 mmHg ) (Active Comparator)
  Interventions: Drug: BP raising drug (phenylephrine) or BP lowering drugs (nicardipine, labetalol, urapidil)

INTERVENTIONS:
Drug: BP lowering drugs (nicardipine, labetalol, urapidil) — After successful reperfusion, appropriate antihypertension medication is administered to control systolic blood pressure <180 mmHg.
  Arms: Conventional BP magnagement group (SBP ≤180 mmHg)
Drug: BP raising drug (phenylephrine) or BP lowering drugs (nicardipine, labetalol, urapidil) — After successful reperfusion, appropriate BP raising (20% increase in SBP, maximum of 160 from baseline SBP) are administered.
  Arms: Intensive BP raising group (20% increase in SBP, maximum of 160 mmHg )

SUMMARY:
Though intravenous thrombolysis has been shown to improve symptoms in acute ischemic stroke patients, the recanalization rate remains low (22.6%) and only around 30% of patients benefit from the treatment. Recently, endovascular thrombectomy using stent retrievers or catheters has proven to be more effective, with a success rate of nearly 80%. However, only 50% of patients experience clinical improvement, highlighting the need for new treatment strategies to enhance outcomes. Current guidelines recommend maintaining systolic blood pressure (BP) below 180 mmHg after thrombectomy, but there is a lack of evidence regarding optimal blood pressure management post-reperfusion.

Four randomized clinical trials, including the OPTIMAL-BP trial, have examined blood pressure control following thrombectomy. Meta-analyses showed that intensive BP lowering did not reduce symptomatic hemorrhage and was associated with worse functional outcomes at 3 months. Specifically, lowering BP too aggressively after successful reperfusion could worsen outcomes by reducing perfusion to the ischemic penumbra. Therefore, this study will investigate whether a more targeted blood pressure elevation strategy could improve patient prognosis compared to standard BP control in those with post-thrombectomy systolic BP below 150 mmHg.

This is a prospective, randomized, open-label trial with blinded endpoint assessment (PROBE) design, aimed at comparing intensive and standard BP control strategies in acute ischemic stroke patients. Participants will be randomized 1:1 into either an intensive BP control group (targeting a 20% systolic BP increase, capped at less than 160 mmHg) or a standard BP control group (systolic BP at or below 180 mmHg).

DETAILED DESCRIPTION:
1. This is a prospective, randomized, open-label trial with blinded endpoint assessment (PROBE) design.
2. Participants will be randomly assigned in a 1:1 ratio to either an intensive BP control group (targeting a 20% increase from baseline systolic BP, capped at less than 160 mmHg) or a standard BP control group (maintaining systolic BP at or below 180 mmHg).
3. Randomization: Allocation will be stratified by stroke severity (NIHSS <15 or ≥15) and participating study center. Randomization will be conducted via a web-based system using a pre-generated randomization table created by a statistician. Investigators will enter stratification variables (study center, NIHSS score) into the system to receive the randomized allocation.
4. This is a multi-center prospective study involving patients admitted to participating hospitals for acute ischemic stroke between October 2024 and December 2029 (last visit date). The study will include patients who undergo successful intra-arterial reperfusion therapy based on current stroke guidelines.
5. Data collection will include the medical history, imaging findings, BP parameters (systolic BP, diastolic BP, BP variability), neurological scores, functional recovery, and quality of life (QoL) measures for eligible participants.
6. Neurological scores, functional recovery, and QoL assessments will be conducted by independent evaluators who are blinded to treatment allocation.
7. All data will be collected using electronic case report forms (e-CRF), and anonymized imaging data will be sent to the coordinating center.
8. The coordinating center will perform blinded quantification of imaging results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* Patients who underwent endovascular thrombectomy for acute ischemic stroke due to large vessel occlusion (ICA, M1, M2, A1, P1, and VBA).
* Successful recanalization of the intracranial artery after endovascular thrombectomy (modified TICI 2b, 2c or TICI 3).
* Patients whose mean systolic blood pressure was measured to be below 150 mmHg on at least two occasions, taken 2 minutes apart, within 2 hours of successful recanalization.

Exclusion Criteria:

* Age <20
* Patients who failed recanalization of the intracranial artery after endovascular thrombectomy (modified TICI ≤ 2a).
* Patients with systolic blood pressure ≥ 150 mmHg after successful recanalization.
* Patients unable to receive antihypertensive medication post-thrombectomy or in whom the investigator believes aggressive blood pressure control could have adverse effects, such as increased risk of hemorrhage.
* Patients who developed symptomatic intracranial hemorrhage before study enrollment, after successful recanalization.
* Patients with pre-existing neurological deficits (modified Rankin Scale, mRS ≥ 3).
* Patients with heart failure with reduced ejection fraction, defined as an ejection fraction <30%.
* Patients with end-stage renal disease requiring renal replacement therapy or chronic kidney disease stage 4 with an estimated glomerular filtration rate (eGFR) <30 mL/min.
* Patients receiving MAO inhibitors.
* Patients who are currently pregnant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2029-12-03 (Estimated); Study Completion 2029-12-03 (Estimated)

PRIMARY OUTCOMES:
Functinal independence | 3 months
  Proportion of patients with a functional independence (defined as mRS ≤ 2) at 3 months, assessed using the modified Rankin Scale (mRS).
Symptomatic Intracranial Hemorrhage (sICH) | 36 hours
  Symptomatic Intracranial Hemorrhage (sICH) after Endovascular Treatment Intracranial hemorrhage or hemorrhagic transformation identified on MRI (GRE or SWI) or CT within 24 ± 12 hours or due to clinical worsening.
  (Symptomatic intracranial hemorrhage is defined according to the European Cooperative Acute Stroke Study III [ECASS III] criteria)
Stroke related death | 3 months
  Stroke related death within 3 months

SECONDARY OUTCOMES:
Shift analysis of mRS score distribution. | 3 months
  Distributional analysis of the modified Rankin Scale (mRS) scores to assess overall functional outcome shift between treatment groups.
NIHSS score at 24 hours after endovascular treatment. | 24 hours
  Difference in National Institutes of Health Stroke Scale (NIHSS) scores between at 24 hours post-EVT.
Major Neurological Improvement at 24 hours, defined as either an NIHSS score of 0-1 or an improvement of 8 or more points. | 3 months
  Proportion of patients achieving substantial neurological recovery within 24 hours after EVT.
Sustained vessel recanalization on CTA/MRA at 24 hours | Discharge and 1 month
  Evaluation of angiographic reperfusion status (modified Thrombolysis in Cerebral Infarction [mTICI] grade ≥2b)
Proportion of functional independence at 1 month. | 3 months
  Percentage of patients achieving mRS 0-2 at 1 month.
Differences in Euro-Q5 instrument. | 36 hours to 1 week
  Differences in scores measured by Euro-Q5 scale.
Incidence of malignant cerebral edema. | 36 hours
  Frequency of radiologically or clinically confirmed malignant cerebral edema after EVT.
Infarction volumes | 36 hours
  Proportion of functional independence according to infarction volumes in DWI
Using intravenous BP lowering drug | 3 months
  Proportion of functional independence according to intrvenous BP lowering drug
Medication induced BP drop | 3 months
  Proportion of functional independence according to medication inuced BP drop
Collateral circulation measured by Tan scale (good collateral is defined as Tan scale 2-3) in baseline CTA. | 3 months
  Proportion of functional independence according to the degree of collateral flow
Variability in blood pressure (e.g., standard deviation, coefficient of variation, VIM, successive variation, and threshold). | 3 months
  Evaluation of outcome associations with multiple BP variability indices
Outcome comparison by baseline ischemic core burden measured with ASPECTS. | 3 months
  Proportion of functional independence according to the ASPECTS (Alberta Stroke Program Early CT Score) on CT or MRI.
Evaluation of differential outcomes in patients who received IV tPA before EVT. | 3 months
  Proportion of functional independence according to prior tPA administration.
Comparison of outcomes according to presence or severity of intracranial atherosclerotic stenosis. | 3 months
  Proportion of functional independence according to intracranial arterial stenosis.
Assessment of outcome differences by number of thrombectomy passes. | 3 months
  Proportion of functional independence according to multiple attempts at endovascular recanalization.
Evaluation of outcomes relative to attainment and timing of post-EVT BP target. | 3 months
  Proportion of functional independence according to achieving the target blood pressure and the time to target on outcomes.
Outcome comparison by initial angiographic reperfusion grade before BP intervention. | 3 months
  Proportion of functional independence according to baseline mTICI scores.
Assessment of outcome differences between patients with and without early neurological worsening. | 3 months
  Proportion of functional independence according to neurological deterioration (NIHSS worsening by ≥4 points).
Evaluation of outcomes stratified by occlusion site (e.g., ICA, M1, M2). | 3 months
  Proportion of functional independence according to the occluded vessel involved.
Biochemical markers including D-dimer, CRP, or glucose | 3 months
  Proportion of functional independence according to laboratory findings including D-dimer, CRP, or glucose.
Evaluation of vascular stiffness as a determinant of post-EVT outcomes. | 3 months
  Proportion of functional independence according to estimated pulse wave velocity (ePWV).
Small artery disease - white matter hyperintensity | 3 months
  Proportion of functional independence according to degree of white matter hyperintensity
Small artery disease - microbleeds | 3 months
  Proportion of functional independence according to number of microbleeds
Small artery disease - old lacunar infarction | 3 months
  Proportion of functional independence according to number of old lacunar infarctions
Optimal target BP according to AI predicting for functional independence in 10 mmHg increments | 3 months
  Model-based identification of the optimal SBP target range predicted by AI for favorable outcomes.
Occurrence of adverse event or serious adverse event | 3 months
  Incidence and type of adverse events
Treatment failure, defined as failure to achieve target blood pressure on two consecutive measurements within 24 hours after endovascular therapy. | 24 hours
  Rate of unsuccessful BP target attainment during the acute post-procedure period.
Differences in BP variability depending on the antihypertensive agent use (labetalol or nicardipine). | 24 hours
  Comparison of short-term BP stability between BP medication used for post-EVT management.
Differences in causes of death. | 3 months
  Comparison of mortality causes
Diffrences in fuctional outcomes at 1 year. | 1 year
  Difference in 1-year functional outcomes according to mRS and EQ-5D-5L.
Euro-Q5-5L analogue scale. | 1 year
  Differnec in scores measured by Euro-Q5 scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After study competition, the participating researcher can submitt the proposal. Publication committee will evaluate the proposal and approve it. After approval, patients data will be shared with researcher.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available until the study was published.